CLINICAL TRIAL: NCT06951802
Title: Endometriosis and Pain Treatment by Intraoperative Administration of Low-dose Ketamine A Single-Centre, Prospective, Randomized, Controlled Trial
Brief Title: Endometriosis and Pain Treatment by Intraoperative Administration of Low-dose Ketamine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-01677
Record Dates: First submitted 2025-04-16; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Ketamine; Propofol

STUDY DESIGN:
Intervention Model Description: Randomised controlled prospective trial in two groups. Group 1 will receive standard anaesthesia with propofol and ketamine. Group 2 will receive standard anaesthesia with propofol alone.
Who Masked: Participant
Masking Description: See description Model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Ketamine (Experimental): Standard anaesthesia with propofol and administration of ketamine.
  Interventions: Drug: Ketamine; Drug: Propofol
- Group Control (Other): Standard anaesthesia with propofol.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ketamine — Low-dose administration of ketamine during laparoscopic surgery
  Arms: Group Ketamine
Drug: Propofol — Control group

SUMMARY:
RCT comparing intraoperative administration of low-dose ketamine during laparoscopic endometriosis operation and the postoperative pain outcome

DETAILED DESCRIPTION:
Endometriosis affects 10% of women of childbearing age and 25% - 50% of infertile women worldwide. Although most patients with endometriosis are completely asymptomatic, there are still a significant proportion of patients whose quality of life is impaired by the disease, resulting in chronic pelvic pain.

Hysterectomy is the most common surgical procedure performed in nonpregnant women when conservative strategies are ineffective. However, there is a poor correlation between objective findings of significant endometriosis and pain severity. Women with endometriosis are at a four-fold greater risk of long-term opioid use than those without endometriosis. Approximately 30% of women who undergo surgery for endometriosis report persistent pain after the surgical removal of the lesion(s). In addition to surgical trauma, other predisposing factors can influence the recovery or progression of chronic diseases, which should be considered when selecting perioperative treatment. Furthermore, studies have shown that in many surgical procedures, incision size and degree of tissue trauma are poorly related to postoperative pain intensity, depending on the pain treatment. After surgery, postoperative pain may be severe overall but usually resolves within the first day of surgery with a Numeric Rating Scale (NRS) pain score ≤ 4. Pain from laparoscopic endometriosis operation includes incisional pain, which may also be severe initially but subsides within the first half of the day; visceral pain that takes longer to resolve (up to a day); and shoulder pain (e.g., shoulder tip pain) that is milder. However, approximately 80% of women develop this condition after gynecologic laparoscopy procedures, which usually disappears within 24 hours and may last for several days. The typical duration of opioid rescue medication use is approximately four days. They should not cause discomfort or limit postoperative recovery.

Although the cause of endometriosis is not yet fully understood, chronic inflammation(s) and increased menstrual bleeding often leads to iron deficiency and even anemia. Iron deficiency anemia is the most common form of anemia, accounting for 50%. In 2019, the prevalence of girls and women of childbearing age (15 - 49 years) with anemia worldwide averaged 30%. For Switzerland, iron deficiency anemia is reported at 11.2 % and is well below the global average. Since iron and its deficiency play an important role in the pathogenesis of endometriosis and possibly also maintain it, it does not surprise that endometriosis patients have an increased risk of iron deficiency or anemia.These patients with a latent or manifest iron deficiency also complain of pain. Up to now, there are only indications that iron could play a role in the proinflammatory pain transmission pathways in endometriosis and could probably maintain and trigger chronic pain. As with nonsurgical chronic pain, psychological and social factors have an important impact that may persist for months or years after surgery. Suboptimal treatment of acute pain has many negative consequences including increased morbidity, impaired physical function and quality of life, slower recovery, prolonged opioid use during and after hospitalization, and increased care costs. Furthermore, in a significant proportion of patients, early postoperative pain appears to trigger pain that may persist for several months. Specifically, younger age, non-white race, lower education, history of sleep disorders, current smoking and alcohol use, high preoperative fibromyalgia screening scores, and high anxiety levels were associated with higher pain severity and excessive pain and may be underlying determinants. Also previous opioid consumption contributes to persistent postoperative pain. As pain is both a sensory and an emotional experience, psychological factors such as mood, disability, and pain coping (e.g., pain self-efficacy and pain catastrophizing) play an important role in this setting. Therefore, patients, particularly those with a predisposition or known tendency for depression, anxiety, or catastrophic symptoms, are at a high risk of developing chronic postsurgical pain. However, in some patients, acute postoperative pain persists beyond the tissue-healing period and develops into a chronic pain state. Approximately 10% of the patients undergoing surgery and 30% of those with endometriosis experience chronic pain. Patients, who have already taken preoperative painkillers or have significantly excessive postoperative analgesic consumption are at a risk of developing chronic pain. Nevertheless, opioids are often overused, particularly during the post discharge period. Even today, acute pain management in the setting of trauma, exacerbation of chronic painful conditions, and postsurgical pain, particularly in patients who are opioid-tolerant remains a challenge in the perioperative setting. In this context, ketamine can be used, generally at subanesthetic doses. However, some patients reported severe debilitating side effects of ketamine administration that did not tolerate higher ketamine doses, an adequate balance of analgesia, and adverse effects in continuous low-dose ketamine in the range of 0.1 - 0.5 mg·kg-1·h-1 was described as sufficient.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for endometriosis operation requiring general anaesthesia at the Inselspital, Bern University Hospital, University of Bern, Department of gynaecology and obstetrics.
* Age ≥ 18 years
* American Society of Anesthesiologist (ASA) physical status 1-3
* Patients with known or suspected endometriosis
* Written informed consent.

Exclusion Criteria:

* Age < 18 years
* ASA physical status ≥4
* Higher-grade atrioventricular block without pacemaker
* Severe hypovolemia or bradycardia
* Uncontrolled hyper- or hypotension
* Liver disease
* Known malignant hyperthermia
* Cardiovascular instability or severe heart failure (New York Heart Association classification (NYHA) > III)
* Myocardial infarction during the last 30 days prior to surgery
* Increased intracranial or increased intraocular pressure
* Limited peripheral autonomic activity, hypersensitivity to ketamine or propofol or its components
* Pregnancy
* Rejection or lack of consent of the patient or relatives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total opioids prescribed and consumed during hospitalization for endometriosis. | During hospitalisation, expected to be on average 2-5 days
  The primary study outcome is the total opioids consumed during hospitalisation (converted in oral morphine equivalents)

SECONDARY OUTCOMES:
Daily pain severity during hospitalization | During hospitalisation, expected to be on average 2-5 days
  Pain score, measured by questionaire, scale from 0 to 10, with higher values corresponding to higher pain level
Postoperative complications | During hospitalisation, expected to be on average 2-5 days
  Number of patients with nausea, vomiting or dizziness
Patient wellbeing | 30 days to 6 months after surgery
  Measured by questionnaire
Preoperative iron status | Preoperatively (expected to be on average 2-5 days prior to surgery)
  Iron status will be classified as normal, latent iron deficiency, or manifest iron deficiency based on laboratory values (e.g., hemoglobin, ferritin, transferrin saturation). Evaluation of manifest or latent iron deficiency, measured by laboratory testing. The scale typically ranges from 0 to over 300 µg/L in clinical practice, but the diagnostic focus is on lower values. For adults, a ferritin concentration below 10-15 µg/L is generally considered indicative of iron deficiency. Higher values indicate better iron stores, but values above the upper reference limit may suggest iron overload or inflammation.
Pain score | During hospitalisation, expected to be on average 2-5 days
  Assessed using the Numeric Rating Scale (NRS), which ranges from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate worse pain. NRS score (0-10)
Total postoperative analgesic consumption before discharge | During hospitalisation, expected to be on average 2-5 days
  The total amount of analgesics consumed postoperatively, converted to intravenous morphine equivalents using standard conversion tables. Higher values indicate greater analgesic requirement. Milligrams of intravenous morphine equivalent (mg IV MEQ)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Vetter, MD, Study Chair — Dep. of Anaesthesiology and Pain Medicine, Inselsptial Bern
Locations (1):
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kanellos P, Nirgianakis K, Siegenthaler F, Vetter C, Mueller MD, Imboden S. Postoperative Pain Is Driven by Preoperative Pain, Not by Endometriosis. J Clin Med. 2021 Oct 15;10(20):4727. doi: 10.3390/jcm10204727. PMID 34682850
- [Background] Abbott J, Hawe J, Hunter D, Holmes M, Finn P, Garry R. Laparoscopic excision of endometriosis: a randomized, placebo-controlled trial. Fertil Steril. 2004 Oct;82(4):878-84. doi: 10.1016/j.fertnstert.2004.03.046. PMID 15482763
- [Background] Chiuve SE, Kilpatrick RD, Hornstein MD, Petruski-Ivleva N, Wegrzyn LR, Dabrowski EC, Velentgas P, Snabes MC, Bateman BT. Chronic opioid use and complication risks in women with endometriosis: A cohort study in US administrative claims. Pharmacoepidemiol Drug Saf. 2021 Jun;30(6):787-796. doi: 10.1002/pds.5209. Epub 2021 Mar 16. PMID 33611812
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Lirk P, Thiry J, Bonnet MP, Joshi GP, Bonnet F; PROSPECT Working Group. Pain management after laparoscopic hysterectomy: systematic review of literature and PROSPECT recommendations. Reg Anesth Pain Med. 2019 Apr;44(4):425-436. doi: 10.1136/rapm-2018-100024. Epub 2019 Feb 3. PMID 30914471
- [Background] Lopez A, Cacoub P, Macdougall IC, Peyrin-Biroulet L. Iron deficiency anaemia. Lancet. 2016 Feb 27;387(10021):907-16. doi: 10.1016/S0140-6736(15)60865-0. Epub 2015 Aug 24. PMID 26314490
- [Background] Cappellini MD, Comin-Colet J, de Francisco A, Dignass A, Doehner W, Lam CS, Macdougall IC, Rogler G, Camaschella C, Kadir R, Kassebaum NJ, Spahn DR, Taher AT, Musallam KM; IRON CORE Group. Iron deficiency across chronic inflammatory conditions: International expert opinion on definition, diagnosis, and management. Am J Hematol. 2017 Oct;92(10):1068-1078. doi: 10.1002/ajh.24820. Epub 2017 Jul 7. PMID 28612425
- [Background] World Health Organization. (2021). Anaemia in women and children. The Global Health Observatory. Retrieved July 4, 2022, from. https://www.who.int/data/gho/data/themes/topics/anaemia_ in_women_and_children
- [Background] Gete DG, Doust J, Mortlock S, Montgomery G, Mishra GD. Risk of Iron Deficiency in Women With Endometriosis: A Population-Based Prospective Cohort Study. Womens Health Issues. 2024 May-Jun;34(3):317-324. doi: 10.1016/j.whi.2024.03.004. Epub 2024 Apr 24. PMID 38658289
- [Background] Maddern J, Grundy L, Castro J, Brierley SM. Pain in Endometriosis. Front Cell Neurosci. 2020 Oct 6;14:590823. doi: 10.3389/fncel.2020.590823. eCollection 2020. PMID 33132854
- [Background] Wyatt J, Fernando SM, Powell SG, Hill CJ, Arshad I, Probert C, Ahmed S, Hapangama DK. The role of iron in the pathogenesis of endometriosis: a systematic review. Hum Reprod Open. 2023 Jul 27;2023(3):hoad033. doi: 10.1093/hropen/hoad033. eCollection 2023. PMID 37638130
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Glare P, Aubrey KR, Myles PS. Transition from acute to chronic pain after surgery. Lancet. 2019 Apr 13;393(10180):1537-1546. doi: 10.1016/S0140-6736(19)30352-6. PMID 30983589
- [Background] Schwenk ES, Viscusi ER, Buvanendran A, Hurley RW, Wasan AD, Narouze S, Bhatia A, Davis FN, Hooten WM, Cohen SP. Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Acute Pain Management From the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists. Reg Anesth Pain Med. 2018 Jul;43(5):456-466. doi: 10.1097/AAP.0000000000000806. PMID 29870457
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB. Fibromyalgia criteria and severity scales for clinical and epidemiological studies: a modification of the ACR Preliminary Diagnostic Criteria for Fibromyalgia. J Rheumatol. 2011 Jun;38(6):1113-22. doi: 10.3899/jrheum.100594. Epub 2011 Feb 1. PMID 21285161
- [Background] Shirvalkar P, Prosky J, Chin G, Ahmadipour P, Sani OG, Desai M, Schmitgen A, Dawes H, Shanechi MM, Starr PA, Chang EF. First-in-human prediction of chronic pain state using intracranial neural biomarkers. Nat Neurosci. 2023 Jun;26(6):1090-1099. doi: 10.1038/s41593-023-01338-z. Epub 2023 May 22. PMID 37217725
- [Derived] Vetter C. Opioid-sparing by low-dose ketamine for endometriosis surgery. A single-center, prospective, randomized, trial. Pain Manag. 2026 Jan 18:1-6. doi: 10.1080/17581869.2026.2613800. Online ahead of print. PMID 41550074